CLINICAL TRIAL: NCT02347475
Title: Impact of Red Cell Transfusion on Superior Mesenteric Artery Flow Patterns and Intestinal Oxygenation in Fed Preterm Neonates (SPARTAN: Sma PAttern Related to TrAnsfusion in Neonates)
Brief Title: SMA Flow Patterns in Neonatal Transfusion
Acronym: SPARTAN
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Amelie Stritzke, MD, University of Calgary
Other Study IDs: 14-0312
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational Study — Ultrasound and NIRS

SUMMARY:
This study aims to measure the changes induced by packed red blood cell (PRBC) transfusion in the superior mesenteric artery (SMA) flow velocity and intestinal oxygenation indices in premature neonates. These changes will be measured in relation to feeding, before and after a blood transfusion. Overall reduction of intestinal perfusion is a risk factor for necrotizing enterocolitis (NEC) - a condition with significant mortality and long term morbidity. Identifying specific patterns of flow velocity and tissue oxygenation changes will allow for planning, studying and implementing risk avoidance and minimization strategies.

DETAILED DESCRIPTION:
Hypothesis: In preterm neonates the anticipated physiologic post-prandial increase in each SMA flow and intestinal perfusion is blunted post transfusion. This is worse in SGA infants and/or in the presence of a PDA.

Questions: 1) Does PRBC transfusion alter postprandial SMA flow increases and intestinal oxygenation indices in preterm infants receiving enteral feeds? 2) Is there a difference in postprandial SMA flow and intestinal perfusion changes in recently transfused SGA infants compared to AGA infants, and in those with and without a PDA? Primary Outcome: Post-prandial SMA flows changes before and after PRBC transfusion.

Secondary outcomes: Pre-post prandial changes in near-infrared spectroscopy (NIRS)-measured intestinal oxygenation parameters before and after PRBC transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity (<34 completed weeks of gestation at birth)
* Need for PRBC transfusion
* Feeding at least 30ml/kg/day at the time of transfusion

Exclusion Criteria:

* Neonates previously diagnosed with gastrointestinal problems such as NEC, intestinal perforation or atresia.
* Infants receiving continuous feeds or less than 30ml/kg/day
* Major congenital or chromosomal abnormalities or infants unlikely to survive
* Skin disruption precluding application of sensors

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prematurity (<34 completed weeks of gestation at birth) Need for PRBC transfusion
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Post-prandial SMA flows changes before and after PRBC transfusion | Just prior to transfusion until 48 hours post completion of transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Stritzke, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada